CLINICAL TRIAL: NCT05589155
Title: Efficacy of Using Mobile Health Applications for Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HS-2022-0156
Record Dates: First submitted 2022-10-16; First posted 2022-10-21 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: diabetes; mhealth; ehealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Healthi (Experimental)
  Interventions: Other: Mobile health application

INTERVENTIONS:
Other: Mobile health application — Intervention will be with mobile health application
  Arms: Healthi

SUMMARY:
The purpose of this study is to determine the effectiveness of mobile health applications in improving health outcomes and type II diabetes outcomes in type 2 diabetics. This study will involve a 6-month long commitment where participants will be expected to weigh themselves every morning, at the same time, and check their blood glucose readings daily before and after meals for at least three meals in the day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type II diabetes for at least 3 months
* Between the age of 18-64
* BMI ≥ 25
* Monitors blood glucose regularly (at least once per day)
* Owns or has access to a bathroom weight scale
* Owns a smartphone and willing to download mobile app

Exclusion Criteria:

* Does not check blood glucose at least once per day
* On medications that promote weight gain such as antipsychotic, antidepressant, and steroid hormone medications.

Medications for diabetes such as insulin, thiazolidinediones or sulfonylureas are oka

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of mHealth apps at changing bodyweight assessed by bodyweight measurements over 6 months | 6 months
  Determine if mhealth app is an effective weight loss modality compared to standard weight loss program (control)
  Outcome measure will be body weight in kg
Self-efficacy in weight management assessed by Weight Management and Nutrition Knowledge questionnaire | 6 months
  Compare and determine which intervention promotes self-efficacy in weight management.
  Reporting will be on a scale of 0-100, with higher scores indicating higher self-efficacy
Long term change in diabetes via A1c | 6 months
  Compare and determine which intervention elicits the most change towards diabetes via HbA1c
  Outcome measure will be HbA1c
Long term change in diabetes via fasting blood glucose | 6 months
  Compare and determine which intervention elicits the most change towards diabetes via fasting blood glucose
  Outcome measure will be fasting blood glucose

SECONDARY OUTCOMES:
Quality of Life after using mHealth apps assessed by World Health Organization Quality of Life BREF questionnaire | 6 months
  Comparing the two arms to determine which leads to greater quality of life (QOL)
  Measures will be reported on a scale of 1-5 across four domains. Scores will be converted to a scale of 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No